## **Study protocol**

## A Multicenter Randomized Trial, Comparing a 25G EUS Fine Needle Aspiration (FNA) Device with a 20G EUS ProCore Fine Needle Biopsy (FNB) Device

**ASPRO trial (ASPiration versus PROcore)** 

ProCore study group

## PROTOCOL TITLE

| Protocol ID | ASPRO trial |
|---|---|
| Short title | Comparing a 25G EUS-FNA with a 20G EUS ProCore |
| | FNB Device |
| Version | Version I |
| Date | 13-10-2014 |
| Coordinating investigator | Drs P.A. van Riet |
| | Department of Gastroenterology & Hepatology, |
| | Room Ca-415, Erasmus University Medical Center, |
| | Rotterdam, the Netherlands |
| | Email; p.vanriet@erasmusmc.nl |
| Principal investigator | Dr D.L. Cahen |
| | Department of Gastroenterology & Hepatology, |
| (See paragraph 3.1 for a list of all | Room H-337, Erasmus University Medical Center, |
| principal investigators per site) | Rotterdam, the Netherlands |
| | Email; djuna@cahen.nl |
| Sponsor | SLO (in Dutch: Stichting Lever Onderzoek, in English: |
| | Foundation for Liver and Gastrointestinal Research) |
| | on behalf of the Department of Gastroenterology and |
| | Hepatology of the Erasmus University Medical Center in |
| | Rotterdam, the Netherlands |
| Subsidising party of | Cook Medical |
| unrestricted grant | O'Halloran Road |
| | National Technology Park |
| | Limerick, Ireland |
| | www.cookmedical.com |
| Independent physician | Dr D. Sprengers |
| | Department of Gastroenterology & Hepatology, Erasmu |
| | University Medical Center, Rotterdam, the Netherlands |

| Laboratory sites | Department of Clinical Pathology, Erasmus University |
|------------------|------------------------------------------------------|
| | Medical Center, Rotterdam, the Netherlands |
| Pharmacy | Not applicable |

## **SUMMARY**

Rationale: During Endoscopic Ultrasound (EUS), tissue samples can be obtained with different techniques. Fine needle aspiration (FNA) provides a cytological specimen. With fine needle biopsy (FNB), a histological specimen is obtained, which generally results in a better diagnostic performance. However, FNB needles are stiffer and more difficult to handle, and can therefore result in less tissue acquisition.

**Objectives**: To compare the performance and diagnostic accuracy of two EUS-guided tissue acquisition devices; a 25G Echotip Ultra Fine Needle Aspiration (FNA) device and a new, more flexible 20G Echotip ProCore Fine Needle Biopsy (FNB) device.

Study design: International randomized multicenter trial.

**Study population:** Patients ≥18 years old, referred for EUS-guided tissue sampling of a: (I) pancreatic mass lesion, (II) lymph node, or (III) other submucosal or undefined mass (non-pancreatic), ≥ I cm in size.

**Intervention:** EUS-guided tissue acquisition by means of either the 25G Echotip Ultra FNA device, or the 20G Echotip ProCore FNB device.

Main study parameters/endpoints: The main endpoint is the diagnostic performance, measured against the *gold standard* diagnosis (based on the surgical resection specimen or in non-operated patients, the outcome of the diagnostic work-up (i.e. tissue sampling and imaging studies), confirmed by a compatible clinical disease course). Secondary endpoints include I. technical success, II, specimen specifics, such as; quality, presence of tissue cores, and pathological classification (cytology, cell-block, or histology), III. procedural aspects, such as; safety, the yield of a single needle pass, and the value of on-site pathological evaluation, and IV. inter-observer variation.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: There are no additional risks involved. Patients are referred for EUS-guided tissue acquisition, as part of the standard diagnostic work-up. Previous reports showed EUS-guided FNA and FNB sampling to be equally safe.